CLINICAL TRIAL: NCT04043013
Title: Influence of Four Different Orthodontic Bracket Prescriptions in Total Posterior Arch Width and Torque Expression
Brief Title: Influence of Four Orthodontic Bracket Prescriptions in Arch Width and Torque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Jose Luis Gandía-Franco, Director, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H1337808714794
Record Dates: First submitted 2019-07-10; First posted 2019-08-02 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Dental Arch Relationship Anomaly
Keywords: ARCH; TORQUE; BRACKET; PRESCRIPTION

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mini-Taurus® (Rocky Mountain©) Brackets (Active Comparator): Brackets Mini-Taurus® (Rocky Mountain©) with:
  ORTHODONTIC BRACKET PRESCRIPTION Canines 0º First Premolar 0º Second Premolar 0º First Molar 0º
  Interventions: Device: Smart Clip® SL3 High Torque (3M Unitek©); Device: Tip-Edge Plus® (TP Orthodontics©); Device: Victory® (3M Unitek©)
- Smart Clip® SL3 High Torque (3M Unitek©) (Active Comparator): Brackets Smart Clip® SL3 High Torque (3M Unitek©) with:
  ORTHODONTIC BRACKET PRESCRIPTION
  Canines +6º First Premolar -4º Second Premolar -4º First Molar -14º
  Interventions: Device: Mini-Taurus® (Rocky Mountain©) Brackets; Device: Tip-Edge Plus® (TP Orthodontics©); Device: Victory® (3M Unitek©)
- Tip-Edge Plus® (TP Orthodontics©) (Active Comparator): Brackets Tip-Edge Plus® (TP Orthodontics©) with:
  ORTHODONTIC BRACKET PRESCRIPTION
  Canines -4º First Premolar -7º Second Premolar -7º First Molar 0º -14º -11º -14º
  Interventions: Device: Mini-Taurus® (Rocky Mountain©) Brackets; Device: Smart Clip® SL3 High Torque (3M Unitek©); Device: Victory® (3M Unitek©)
- Victory® (3M Unitek©) (Active Comparator): Brackets Victory® (3M Unitek©) with:
  ORTHODONTIC BRACKET PRESCRIPTION
  Canines 0º First Premolar -7º Second Premolar -7º First Molar -14º
  Interventions: Device: Mini-Taurus® (Rocky Mountain©) Brackets; Device: Smart Clip® SL3 High Torque (3M Unitek©); Device: Tip-Edge Plus® (TP Orthodontics©)

INTERVENTIONS:
Device: Mini-Taurus® (Rocky Mountain©) Brackets
  Arms: Smart Clip® SL3 High Torque (3M Unitek©); Tip-Edge Plus® (TP Orthodontics©); Victory® (3M Unitek©)
Device: Smart Clip® SL3 High Torque (3M Unitek©)
  Arms: Mini-Taurus® (Rocky Mountain©) Brackets; Tip-Edge Plus® (TP Orthodontics©); Victory® (3M Unitek©)
Device: Tip-Edge Plus® (TP Orthodontics©)
  Arms: Mini-Taurus® (Rocky Mountain©) Brackets; Smart Clip® SL3 High Torque (3M Unitek©); Victory® (3M Unitek©)
Device: Victory® (3M Unitek©)
  Arms: Mini-Taurus® (Rocky Mountain©) Brackets; Smart Clip® SL3 High Torque (3M Unitek©); Tip-Edge Plus® (TP Orthodontics©)

SUMMARY:
The study compares torque and arch width changes between four different orthodontic bracket prescriptions and determine whether changes in dental torque are correlated to changes in arch width at the end of orthodontic treatment.

From an initial sample of 250 patients who sought treatment at the Department of Orthodontics (University of Valencia, Spain), a subsample of 76 patients (31 men and 45 women) were selected to meet inclusion criteria.

The sample was randomly allocated into four groups according to four different orthodontic bracket prescriptions: Prescription A (n=22): Mini-Taurus® (Rocky Mountain©); Prescription B (n=17): Smart Clip® SL3 High Torque (3M Unitek©); Prescription C (n=18): Tip-Edge Plus® (TP Orthodontics©); Prescription D (n=19): Victory® (3M Unitek©).

Initial (T0) and final (T1) plaster and digital study models were available for all patients. Measurements were taken from frontal and occlusal images of the models by a single experienced operator.

DETAILED DESCRIPTION:
Subjects Seventy-six patients (31 men and 45 women) were recruited to participate in the clinical study and who fulfilled the inclusion and exclusion criteria. The inclusion criteria were: Presence of permanent dentition from the first permanent molar, from one side to the other, absence of anomalies in number, size and dental shape, no pre-treatment transversal discrepancies, equivalency in pre-treatment vertical relationships, good quality of study models, no medical contra-indications to the use of fixed appliances and good standard of oral hygiene.

The exclusion criteria were: Presence of oral habits. need to use of two band expansive appliances through the treatment, need of an orthodontic treatment with extractions or requiring orthognathic surgery as a part of their treatment. Subject age and gender were not taken as exclusion criteria, as these variables were not expected to influence the research outcomes.

Sample size calculation A pre-study sample size calculation was performed; power analysis showed that a sample size of at least 64 patients would provide an 80% probability of detecting a medium effect (f=0.2) associated with the interaction term, using an ANOVA model at a confidence level of 95% and assuming a correlation among repeated measurements of 0.5.

Study design: Orthodontic prescription techniques Subjects were chosen randomly and prospectively. Using sealed envelopes with the letters A to D, which corresponded to the 4 treatment groups, patients were parallelly randomly allocated according to the orthodontic bracket prescription of each particular technique so that patients each received either Prescription A (n=22): Mini-Taurus (Rocky Mountain); Prescription B (n=17): Smart Clip SL3 High Torque (3M Unitek); Prescription C (n=18): Tip-Edge Plus (TP Orthodontics); and Prescription D (n=19): Victory (3M Unitek). All underwent standard orthodontic treatments with good occlusal results.

Blinding Once the patient had been randomly allocated to one group or another, it was not possible to blind either the patient or the operator to the bracket type.

Settings All brackets had 0.22 inch slots. Since arch width is directly related to archwire form, the same arch form was used for all 4 techniques: Ovoid Arch FormOrthoForm III (3M Unitek). All patients followed the same archwire sequence starting with a 0.012 SE NiTi (superelastic niquel titanium) archwire, followed by a 0.016 SE NiTi, 0.016 x 0.025 SE NiTi and a 0.019 x 0.025 SE NiTi. The last wire used was a 0.019 x 0.025 inch stainless steel archwire. Two operators (C.G and N.Z) with the same background and experience treated the patients. The arch form was not modified during treatment by either expansion or contraction of the archwires. In all cases, stainless steel ligatures were used, except in technique C where the self-ligating system was applied.

Measurements Occlusal and frontal digital models corresponding to all subjects' upper arches were taken from the initial and final plaster study models. Models were digitalized using the iTero Element digital scanning system. All the models were digitalized by the same operator under identical light conditions.

All measurements were carried out by the same operator (B.T) using the Orthocad software. The operator registered the measurements as T0 (pre-treatment values) and T1 (post-treatment values).

Occlusal images were used to measure intercanine, interpremolar and intermolar widths (mm) from initial (T0) and final (T1) study models. A specific protocol was used to take the following interarch width measurements before and after treatment:

Intercanine width: distance between the cusp tips of bilateral canines. First interpremolar width: distance between the vestibular cusp tips of first bilateral premolars.

Second interpremolar width: distance between the vestibular cusp tips of second bilateral premolars.

Intermolar width: distance between mesiovestibular cusps of first bilateral molars.

Frontal images were used for measuring torque (º) of bilateral canines, first premolars, second premolars, and molars from initial (T0) and final (T1) study models. The torque of maxillary arches was measured before (T0) and after (T1) treatment.

Measurements were taken on the basis of:

Reference lines: two reference lines were established.

1. Horizontal line: line passing through the mesiovestibular cusps of right and left first superior molars.
2. Vertical line: perpendicular to the former line, passing through the centre of the papilla between the two superior central incisors.

Crown axis lines: parallel lines to the vestibular contour of the crowns of canines, premolars and molars, running from the vestibular cusp to the highest point of the gingival margin visible from the frontal projection.

Torque measurements: The angle between the vertical line and the crown axis line of each tooth. Torque was measured and given a positive, negative or 0º value. Positive or negative values were assigned based on the clockwise or counterclockwise divergence of the lines, whereas a 0º value was assigned when they were parallel.

Depending on the torque values at T0, variations in torque at T1 were classified as follows:

Negative torque value: when higher negative values were measured at T0 than T1 (e.g. -5º at T0 and -2º at T1).

Positive torque value: when higher positive values were measured at T0 than T1 (e.g. 5º at T0 and 2º at T1).

ELIGIBILITY:
Inclusion Criteria:

* Presence of permanent dentition from the first permanent molar, from one side to the other.
* Absence of anomalies in number, size and dental shape
* No pre-treatment transversal discrepancies
* Equivalency in pre-treatment vertical relationships
* Good quality of study models
* No medical contra-indications to the use of fixed appliances
* Good standard of oral hygiene

Exclusion Criteria:

* Presence of oral habits
* Need to use of two band expansive appliances through the treatment
* Need of an orthodontic treatment with extractions
* Requiring orthognathic surgery as a part of their treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Change of posterior torque from the initial occlusion to the final occlusion at the end of the orthodontic treatment. | Measurement 1: At the begining of orthodontic treatment. Measurement 2: through orthodontic treatment completion, an average of 18 months
  Degrees
Change of arch width from the initial occlusion to the final occlusion at the | Measurement 1: At the beginning of orthodontic treatment. Measurement 2: through orthodontic treatment completion, an average of 18 months
  Millimeters

IPD SHARING:
Plan to Share IPD: No